CLINICAL TRIAL: NCT06457633
Title: Effectiveness of Experiential Fibrowalk Therapy for Fibromyalgia Based on Pain Science Education, Exercise Therapy, Psychological Support, and Nature Exposure: A Pragmatic Randomized Controlled Trial
Brief Title: Effectiveness of Experiential Fibrowalk Therapy
Acronym: EFW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Experiential Fibrowalk
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Multicomponent Treatment; Nature therapy; Mindfulness; Physical therapy; Pain Science Education (PSE); Psychological Approach; Experiential Therapy
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Single-blind, parallel-group, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experiential FW (Experimental): Group treatment protocol of 12 weekly 120 minute sessions (outdoor intervention) based in no-responder predictive analysis and co-creating process
  Interventions: Behavioral: Experiential FW
- Traditional FW (Active Comparator): Group treatment protocol of 12 weekly 120 minute sessions (outdoor intervention)
  Interventions: Behavioral: Traditional FW
- Online FW (Active Comparator): Group treatment protocol of 12 weekly 60 minute sessions (virtual intervention)
  Interventions: Behavioral: Online FW

INTERVENTIONS:
Behavioral: Experiential FW — Traditional Fibrowalk based on Pain Science Education (30 min.) - Cognitive restructuring (30 min.) - Mindfulness techniques (30 min.) - Physical exercise in a natural environment / nature exposure (30 min.) carried out experientially.
  Arms: Experiential FW
Behavioral: Traditional FW — Traditional Fibrowalk based on Pain Science Education (30 min.) - Cognitive restructuring (30 min.) - Mindfulness techniques (30 min.) - Physical exercise in a natural environment / nature exposure (30 min.)
  Arms: Traditional FW
Behavioral: Online FW — Traditional Fibrowalk based on Pain Science Education (30 min.) - Cognitive restructuring (30 min.) - Mindfulness techniques (30 min.) - Physical exercise in a natural environment / nature exposure (30 min.) performed virtually.
  Arms: Online FW

SUMMARY:
The present project will evaluate through a randomised controlled clinical trial with 4-month follow-up, the efficacy in clinical symptoms and quality of life (3-month time horizon) of the multicomponent EXPERIENTIAL FIBROWALK programme in treating individuals diagnosed with fibromyalgia, in compare with original Fibrowalk and virtual Fibrowalk. Pre-post changes will be evaluated in various variables under investigation, will include kinesiophobia, physical function, anxiety, depression, physical dysfunction, overall impact, and symptom intensity.

The design of the present study with 3 treatment branches:

Condition or disease Fibromyalgia Intervention/treatment Behavioral: TAU + Experiential Fibrowalk Behavioral: TAU + Fibrowalk Behavioral: TAU + virtual

DETAILED DESCRIPTION:
The objective of the Experiential Fibrolwalk study is to determine the clinical effectiveness of a new treatment protocol for individuals with fibromyalgia. This protocol was developed by identifying predictors of poor response and through collaboration between physiotherapists, clinical psychologists, and patients. The objectives of this 4-month controlled clinical trial are twofold. Firstly, it aims to assess the impact of a protocol developed collaboratively by clinical therapists and users on the quality of life of individuals with fibromyalgia. Secondly, it aims to determine the pre-post changes in kinesiophobia, physical function, anxiety, depression, physical dysfunction, overall impact, and symptom intensity. Methods and analysis: The study will involve 120 fibromyalgia patients recruited from the Central Sensitivity Syndromes Specialized Unit at Vall d'Hebron Hospital's Rheumatology Service, who will be randomly assigned to one of three study groups: TAU + Experiential Fibrowalk, TAU + Fibrowalk, TAU + virtual. A comprehensive assessment to collect functional impact, depressive-anxiety symptoms, physical function, fatigue, kinesiophobia, pain catastrophism, impression of change,quality of life variables will be conducted pre-intervention, at half of the intervention (6 weeks), post-intervention (12 weeks), and at 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 to 75 years-old.
* 1990 American College of Rheumatology (ACR) classification criteria + the 2011 modified ACR diagnostic criteria for fibromyalgia
* Able to understand Spanish and accept to participate in the study.

Exclusion Criteria:

* Participating in concurrent or past RCTs (previous year).
* Comorbidity with severe mental disorders (i.e. psychosis) or neurodegenerative diseases (i.e. Alzheimer) that that would limit the ability of the patient to participate in the RCT.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQR) | Change from baseline values at 3 months
  Standard pharmacological treatment usually provided to patients with fibromyalgia. The FIQR comprises three dimensions: physical dysfunction (scores from 0 to 30), overall impact (scores from 0 to 20), and intensity of the symptoms (scores from 0 to 50) is used to measure the impact generated by FM during the last week. It consists of 21 items, which are answered on a numerical rating scale of 11 points (from 0 to 10). Total scores can range from 0 to 100, with higher scores reflecting greater deterioration.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Change from baseline values at 3 months
  HADS is used to quantify the severity of anxiety and depression symptoms. It consists of two dimensions (anxiety and depression) of 7 items each responding on a Likert scale of 4 points. Total scores of each scale (HADS-A and HADSD) range from 0 to 21, where higher scores indicate greater severity of symptoms
Short Form-36 Health Survey (SF-36) | Change from baseline values at 3 months
  Physical Function of the 36-Item Short Form Survey (SF-36) was used to measure physical function. This dimension comprises a total of 10 items, which are answered on a Likert scale of 3 points. Total scores on each scale are then transformed and can range from 0 to 100, with higher scores indicate better physical function.
Tampa Scale for kinesiophobia (TSK-11) | Change from baseline values at 3 months
  TSK-11 is used to assess fear of pain and movement. It consists of 11 items, which are answered on a Likert scale of 4 points. Total scores of each scale range from 11 to 44, where higher scores indicate a greater fear of pain and Movement.
Multidimensional Fatigue Inventory (MFI) | Change from baseline values at 3 months
  Change from baseline values at 6 months] MFI is used to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue. Its consists in a 20-item scale designed. Participants utilize a 7-point scale to express the extent to which specific statements accurately reflect their fatigue experiences. Several positively phrased items are reverse-scored. Greater overall scores indicate higher levels of fatigue severity.
Pain Catastrophising Scale (PCS) | Change from baseline values at 3 months
  PCS is used to evaluate catastrophic thoughts associated with pain. It consists of three dimensions (rumination, magnification, and helplessness) of 13 items in total, which are answered on a Likert scale of 5 points. Total scores on each scale range from 0 to 52, with higher scores indicating more catastrophic thoughts
Psychological inflexibility in pain scale (PIPS) | Change from baseline values at 3 months
  A 12-item scale that assesses psychological inflexibility in pain patients and includes two factors: avoidance and cognitive fusion with pain. Respondents are asked to rate items on a 7-point scale that ranges from 1 (never true) to 7 (always true). Higher scores indicate greater levels of psychological inflexibility.
The Patient Global Impression of Change (PGIC) | Change from baseline values at 3 months
  Is a measure that has been frequently used as indicators of meaningful overall change [on a 7-point Likert scale, from 1 = "Much better" to 7 = "Much worse"] in treatments for chronic pain.
Pain Specific Impression of Change (PSIC) | Change from baseline values at 3 months
  The PSIC asks about the impression of change in more specific domains than PGIC: physical and social functioning, work-related activities, mood, and pain [on a 7-point Likert scale, from 1 = "Much better" to 7 = "Much worse"].
Credibility/Expectancy Questionnaire (CEQ) (Adapted version) | Change from baseline values at 3 months
  This is a 6-item test used to assess treatment expectations (3 items) as well as credibility (3 items). After the treatment, the test is administered with the questions reformulated in the past tense.
Adverse effects of treatments | Change from baseline values at 3 months
  Ad hoc measure to check for the presence of negative effects of psychological treatments.
Socio-demographic questionnaire | Change from baseline values at 3 months
  Gender, date of birth, marital status, living arrangements, educational level and employment status.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Feliu, PhD, Study Chair — Universitat Autonoma de Barcelona
Locations (1):
- Hospital Universitari Vall d'Hebron Research Institute, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No